CLINICAL TRIAL: NCT03719300
Title: A Phase 2 Study of BC-819 in Patients With Non-Muscle Invasive Bladder Cancer Whose Disease is Unresponsive to Bacillus Calmette-Guerin
Brief Title: Codex: Study of Inodiftagene Vixteplasmid (BC-819) in Unresponsive NMIBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Anchiano Therapeutics Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-819-18-204
Record Dates: First submitted 2018-10-18; First posted 2018-10-25 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
Keywords: BCG-unresponsive
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm BC-819 (Experimental): inodiftagene vixteplasmid
  Interventions: Drug: inodiftagene vixteplasmid

INTERVENTIONS:
Drug: inodiftagene vixteplasmid — BC-819 at 20 mg/50 mL, instilled intravesically into the bladder, with a retention time of at least 30 minutes (up to 2 hours).
  Induction Phase (weekly treatments): 10 weekly treatments; Maintenance Phase: treatment every 3 weeks for up to 84 additional weeks
  Other Names: BC-819

SUMMARY:
This study, BC-819-18-204, is a Phase 2, open-label, monotherapy, single-arm, multicenter clinical trial of BC-819 (inodiftagene vixteplasmid) in patients with NMIBC adequately treated with Bacillus Calmette-Guerin (BCG) whose disease is BCG unresponsive according to the US Food and Drug Administration (FDA) guidance.

DETAILED DESCRIPTION:
BC-819 (inodiftagene vixteplasmid) is a recombinant DNA plasmid that directs the expression of a potent toxin specifically in malignant cells but not in normal tissue. It has been designed to exploit the established biology of the H19 gene, which is upregulated and expressed at high levels only in malignant cells, to produce bacterial diphtheria toxin only in bladder cancer tissue. BC-819 is administered directly into the bladder to enable maximal topical exposure to target bladder cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age at the time of consent
2. Patient must have been adequately treated with BCG defined as at least one of the following (FDA 2018):

   1. At least five of six doses of an initial induction course plus at least two of three doses of maintenance therapy
   2. At least five of six doses of an initial induction course plus at least two of six doses of a second induction course
   3. A single course of induction BCG can qualify if the patient has T1 high-grade disease at first evaluation (see 3c)
3. Patient must be BCG-unresponsive defined as at least one of the following (FDA 2018):

   1. Persistent or recurrent CIS alone or with recurrent Ta/T1 disease within 12 months of completion of adequate BCG therapy. An assessment within 15 months can also qualify when no assessment was done 12 months after completion of adequate BCG therapy.
   2. Recurrent high-grade Ta/T1 disease within 6 months of completion of adequate BCG therapy. An assessment within 9 months can also qualify when no assessment was done 6 months after completion of adequate BCG therapy.
   3. T1 high-grade disease at the first evaluation following a single course of induction BCG qualifies (Lerner et al. 2015, Steinberg et al. 2016)
4. Patient must have, at study entry, NMIBC indicated by 1 or more of the following:

   1. Ta or T1 high-grade disease
   2. CIS disease
5. Patient must have no known evidence of concomitant upper tract urothelial carcinoma or urothelial carcinoma within the prostatic urethra within 6 months of enrollment
6. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2
7. Patient must have adequate hematologic function, as demonstrated by the following:

   1. Hemoglobin level ≥10 g/dL
   2. Absolute neutrophil count ≥1.5 x 109/L
   3. Platelet count ≥100 x 109/L
8. Patient must have adequate liver and renal function as demonstrated by the following:

   1. Aspartate aminotransferase and alanine aminotransferase each ≤3.0 x upper limit of normal
   2. Total bilirubin ≤1.5 x upper limit of normal, unless prior documentation of Gilbert's syndrome in which case, 3.0 mg/dL is allowed
   3. Serum creatinine ≤1.5 x upper limit of normal or measured or calculated creatinine clearance ≥30 mL/min
9. Female patients of childbearing potential must use maximally effective birth control during the period of therapy and for 1 month after the last study drug infusion
10. Male patients who are sexually active must be willing to use a double barrier contraceptive method upon study enrollment, during the course of the study, and for 1 month after the last study drug infusion

Exclusion Criteria:

1. Patient has current or previous evidence of muscle invasive (muscularis propria) or metastatic bladder cancer disease
2. Patient has received prior investigational therapy for NMIBC
3. Patient has received any therapy for NMIBC within 10 weeks before the start of study treatment other than surgical resection, 1 dose of chemotherapy, and previous BCG
4. Patient is intolerant to previous BCG treatment in the absence of meeting other criteria for BCG unresponsiveness and adequate BCG therapy
5. Patient has received external beam radiation therapy for bladder cancer at any time or for any other condition
6. Patient has an active infection, including urinary tract infection (viral, bacterial, or fungal) and cystitis
7. Patient has urinary tract signs or symptoms that preclude retention of drug in the bladder; this does not include anticholinergic drugs
8. Patient is known to have tested positive for human immunodeficiency virus (HIV). No HIV testing is required if patient is not known have tested positive
9. Patient is female and is pregnant or breastfeeding
10. Patient has a known presence or history of malignancy of other organ system within the 5 years before study start, with the exception of non-melanoma skin cancer; very low or low-risk prostate cancer; or patients who have been disease free for at least 2 years following stage 1 or 2 cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Alaska Urological Institute, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - American Institute of Research, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - The Urology Center of Colorado, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Florida Health Jacksonville, Shands Hospital, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - University of Illinois Hospital and Health Systems (Outpatient Care Center), Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Wichita Urology Group, Wichita, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Clinical Foundation, New Orleans, Louisiana
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - New Jersey Urology, LLC, Belleville, New Jersey
  - MD Anderson Cancer Center at Cooper, Voorhees Township, New Jersey
  - Albany Medical College, Albany, New York
  - Weill Cornell Medical College - NY Presbyterian Hospital, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Chapel Hill Hospital, Urology Clinic, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - Carolina Urology Partners, PLLC, Huntersville, North Carolina
  - University of Toledo, Dept. of Urology and Kidney Transplant, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University South Carolina, Charleston, South Carolina
  - Regional Urology, Greenville, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - The Methodist Hospital d/b/a Houston Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - West Virginia University Cancer Institute, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were patients with High Risk Non Muscle Invasive Bladder Cancer whose disease was unresponsive to BCG. It was planned to enroll and treat 140 patients (N=140), of which 70 to 100 were estimated to have carcinoma in situ (CIS) (with or without papillary disease).
Groups:
- Single Arm BC-819: The administration of BC-819 was separated into 2 phases, the induction phase, and the maintenance phase. During the induction phase, patients were to receive an intravesical instillation of BC-819 at a dose of 20 mg/50 mL aqueous solution once per week for 10 weeks according to the induction phase treatment schedule. Upon completion of the induction phase, patients transitioned to maintenance therapy of BC-819 every 3 weeks beginning at Week 12 (Visit 11) and continuing for the next 84 additional weeks until the end of the study, defined as completion of the 96-week visit (Visit 39).
Period: Overall Study
Arm/Group | Single Arm BC-819
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 72.3 [57 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 104.4 (36.8)
Height [Mean (Standard Deviation); unit: cm] | 172.0 (21.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 39.7 (36.5)
Baseline ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status is used by healthcare professionals to assess the progression of disease in cancer patients and is a standard criteria to determine how the disease impacts patient's daily living abilities.
  GRADE ECOG PERFORMANCE STATUS
  0 Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light nature.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities
  3. Capable of only limited selfcare
  4. Completely disabled
  5. Dead
  Participants
    0: Fully active | 30
    1: Restricted activity but ambulatory | 0
    2: Ambulatory | 2

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Baseline CIS That Achieve a Complete Response After Treatment With BC-819 (Measured at 12 Weeks)
Description: Complete response is defined as at least one of the following:
  * Negative cystoscopy and negative (including atypical) urine cytology
  * Positive cystoscopy with biopsy-proven benign or low-grade NMIBC and negative cytology
  * Negative cystoscopy with malignant urine cytology if cancer is found in the upper tract or prostatic urethra and random bladder biopsies are negative
  The complete response in patients with CIS for this endpoint was documented on or after the Week 12 response assessment and on or prior to the Week 48 assessment. Duration of complete response in patients with CIS was calculated from the documented onset of the complete response to the assessment where the patient no longer met the definition of complete response.
Time Frame: 12 weeks
Population: 17 participants had efficacy assessment for this Outcome Measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 17
Percentage of participants | 17.6 [3.8 to 43.4]

2. Secondary Outcome: Percentage of Patients With Absence of High-grade Recurrent or Persistent Disease at 48 Weeks (Overall Population and Subgroup of Patients With CIS)
Description: Time to recurrence (Kaplan-Meier plot) recurrence is defined as the reappearance or persistence of high-grade disease, or new high-grade disease. Recurrence must be biopsy proven. Persistence, appearance, or presence of lower grade disease was not considered to be a recurrence event
Time Frame: 48 weeks
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Patients With Absence of High-grade Recurrent or Persistent Disease at 12, 24, 36, 72, and 96 Weeks (Overall Population and Subgroup of Patients With CIS)
Description: as for outcome 2
Time Frame: 12, 24, 36, 72, and 96 weeks
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Patients Who Are Progression-free at 48, 72, and 96 Weeks
Description: The incidence of PFS at 48, 72, and 96 weeks as well as time to progression estimated using Kaplan-Meir methods. Progression is defined as the development of T2 or greater disease. Sensitivity analyses was performed and included any of the following as progressions:
  * An increase in stage from Ta or CIS to T1, or
  * Development of T2 or greater, or
  * Lymph node disease, or
  * Distant metastasis
Time Frame: 48, 72, and 96 weeks
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival of Patients Enrolled in the Study at 48, 72, and 96 Weeks
Description: Overall survival of patients enrolled in the study at 48, 72, and 96 weeks and survival time was estimated using Kaplan-Meier methods
Time Frame: 48, 72, and 96 weeks
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life in Patients Treated With BC-819
Description: Measured by the The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30), a general questionnaire for assessing quality of life in cancer patients, and the Non-Muscle Invasive Bladder Cancer Questionnaire (QLQ-NMIBC24 ) for patients with NBIMC disease. EORTC QLQ-C30 include five functional scales , three symptom scales, a global health status/quality of life scale, and six single items. QLQ-NMIBC24 include five multi-item symptom scales, one multi-item functional scale, and five single-item measures.These scales range in score 0-100 scale and an for functional scales, a higher a higher score corresponds to greater function or quality of life. For symptom scales, a higher score corresponds to greater symptom burden.
Time Frame: 48, 72, and 96 weeks
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

7. Secondary Outcome: Assessment of Safety
Description: The safety was evaluated by assessment of AEs according to CTCAE version 5.0, regardless of relationship to study medication.
Time Frame: 9 months
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to Recurrence (Kaplan-Meier Plot)
Description: as for outcome 2
Time Frame: 12, 24, 36, 72, and 96 weeks
Population: Data were not collected.
Arm/Group | Single Arm BC-819
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Single Arm BC-819
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm BC-819 (N=32)
Acute left ventricular failure (Cardiac disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm BC-819 (N=32)
Diarrhoea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Chills (General disorders) | 2
Urinary Tract Infection (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Micturition urgency (Renal and urinary disorders) | 7
Dysuria (Renal and urinary disorders) | 6
Pollakiuria (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 3
Bladder spasm (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03719300/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03719300/SAP_001.pdf